CLINICAL TRIAL: NCT00018135
Title: Parathyroid Hormone Levels in Relation to the Phosphorus Content of Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Prevention
Other Study IDs: NCRR-M01RR00036-0795
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Renal Failure
Keywords: high iPTH levels
MeSH Terms: conditions — Renal Insufficiency | interventions — calcium acetate; Aluminum Hydroxide; Sevelamer

INTERVENTIONS:
Drug: calcium acetate
Drug: aluminum hydroxide
Drug: Sevelamer

SUMMARY:
Patients on hemodialysis tend to have chronic elevations in the level of phosphorus in the blood and a secondary increase in the iPTH level. This chronic elevation in iPTH can have adverse consequences, thus a variety of phosphate binders are given in an attempt to decrease the absorption of phosphorus present in the normal diet. Some preliminary studies have indicated that the iPTH level may change based on the amount of phosphorus present in a meal prior to any significant absorption of phosphorus. If this is true in hemodialysis patients, then the timing of the administration of phosphate binders in relation to the ingestion of meals needs to be considered

DETAILED DESCRIPTION:
Drugs used will include three phosphate binders already approved and commonly used. Calcium acetate, aluminum hydroxide, and sevelamer (Renagel) will be given on separate occasions in conjunction with a high phosphorus meal. They will be given in standard doses used in the treatment of high phosphorus levels in hemodialysis patients.

The population targeted will included hemodialysis patients with elevated iPTH and phosphorus levels.

The patients will receive up to five separate meals. Four of these will be high phosphorus content meals and one will be a low phosphorus content meal. On up to three occasions with the high phosphorus content meals the patients will ingest one of the three phosphate binders. The meals will be ingested after a twelve-hour overnight fast. Labs will be drawn prior to meal ingestion and then at 15, 30, 60, 120 and 240-minute intervals. The labs will consist of iPTH, phosphorus, calcium, and glucose. A serum albumin level will be obtained with the initial specimen only. The patients will have an iPTH level of at least 200pg/ml and a serum phosphorus level of at least 4.0 mg/dl.

The primary outcome will be the change in the iPTH level in relation to the phosphorus content of the meals. Secondary outcomes will include the change in iPTH level in relation to the various phosphate binders being used.

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years of age or older
* Receiving treatment with hemodialysis for at least 90 days
* Serum iPTH levels greater than 200pg/ml
* Serum phosphorus levels greater than 4.0mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086